CLINICAL TRIAL: NCT05166278
Title: The Effectiveness of Verbal and Non-verbal De-escalation Techniques on Reduction of Aggressive Behaviour and Coercion
Brief Title: The Effectiveness of De-escalation in Management of Aggression
Acronym: EDtAC_AC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Centre Maribor (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRP-2018/01-09
Record Dates: First submitted 2021-12-14; First posted 2021-12-21 (Actual); Last update posted 2021-12-21 (Actual); Status verified 2021-12

CONDITIONS: Aggression; Physical Restraint; Education
Keywords: aggression; coercion; physical restraint; de-escalation training; intervention; effectiveness
MeSH Terms: conditions — Aggression | interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: During the five months of the baseline period, the management of aggressive behavior in all psychiatric hospitals will be the same as usual. Before the five months of the intervention period, hospitals will be randomly assigned to either an experimental or control group in the 1:1 ratio. The staff in the experimental group will receive training in verbal and nonverbal de-escalation techniques, and in the control group, the staff will manage aggressive behavior as usual. Regular annual training on the use of coercive measures will be conducted as usual in all hospitals during the study.
Who Masked: Outcomes Assessor
Masking Description: The hospital staff will be unaware of the aim and the design of the study. All psychiatric hospitals will be informed that de-escalation training will be provided within 2 years.
  Data from the SOAS-R forms and documentation for the use of physical restraint will be transferred to electronic databases by an independent collaborator who is not familiar with the design of the study. The randomization will be performed after the baseline period, so the baseline data could not be biased.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EXPER (Experimental): Deescalation training.
  Interventions: Behavioral: De-escalation training
- CONTR (No Intervention): Management of aggressive behaviour as usual.

INTERVENTIONS:
Behavioral: De-escalation training — The intervention will include training on verbal and nonverbal de-escalation techniques. The training will be prepared according to the recommendations of the Beta Project of the American Association for Emergency Psychiatry, the World Health Organization Quality Rights training to act, unite and empower for mental health and a handbook for the use of de-escalation skills in a hospital setting by Amdur E. The first part of the education is based on theoretical backgrounds: aggressive behavior in a psychiatric patient, risk factors, focusing on factors that can be modified, communication, de-escalation. The second part is a practical workshop. The training will be 16 hour duration in total. A short handbook and a list of verbal and non-verbal approaches will be prepared for all staff members involved in the training.
  Other Names: Education
  Arms: EXPER

SUMMARY:
A multicenter, intervention study will be conducted in all psychiatric hospitals in Slovenia.

The purpose of the study is to evaluate the effect of verbal and non-verbal de-escalation techniques on the incidence and severity of aggressive behavior and on the incidence and duration of physical restraints. The proposed hypothesis is that de-escalation training and regular use of de-escalation can reduce aggressive incidents and the use of physical restraints in the acute psychiatric ward.

In Slovenia, inpatient psychiatric treatment is provided by six psychiatric hospitals. There are two acute psychiatric wards in each hospital, one for male and one for female patients. All hospitals will be invited to participate in the study.

The study will be carried out in two phases, a baseline period of five consecutive months and an intervention period of the same five consecutive months in the following year. At the end of the baseline period, hospitals will be randomly assigned to either the experimental or control group.

The intervention will include training on verbal and nonverbal de-escalation techniques for staff teams in experimental wards. The first part of the education is based on theoretical backgrounds: aggressive behavior in a psychiatric patient, risk factors, communication, de-escalation. The second part is a practical workshop. The training will be 16-hour duration in total. A short handbook and a list of verbal and non-verbal approaches will be prepared for all staff members involved in the training.

For the baseline and intervention phase, data on the number and severity of aggressive incidents, the number and duration of physical restraint episodes, and the number of aggressive or restrained patients will be obtained.

DETAILED DESCRIPTION:
Aggression is a serious problem in acute psychiatric settings, often followed using physical restraints. Guidelines for the management of aggressive behavior recommend the use of de-escalation techniques as the first choice but evidence of their effectiveness is still limited. Aggression management studies often involve several organizational and structural interventions in the ward environment, staff, and patient management, which can be expensive and time consuming. Two Cochrane reviews (Du M et al. 2017, Spencer S et al. 2018) revealed a lack of relevant studies on the effectiveness of de-escalation techniques in managing aggression. The method of measuring the impact of de-escalation is often assessing the frequency of coercive measures, especially physical restraints. A significant proportion of physical restraints are not a consequence of aggression, so it is important to monitor aggressive incidents and physical restraints according to the reason for the application.

This research will be carried out within the National project of Slovenian Psychiatric Association, aimed to reducing aggressive behavior and the use of coercive measures in acute psychiatric units. Following visits by the CPT's (European Committee for the Prevention of Torture and Inhuman or Degrading Treatment or Punishment) to Slovenian psychiatric hospitals with recommendations for greater emphasis on the use of de-escalation before the introduction of coercive measures, a decision was made to prepare de-escalation training for all psychiatric hospitals. During this project, we will conduct the research to evaluate the effectiveness of de-escalation on the incidence and severity of aggressive behavior and on the incidence and duration of physical restraints due to aggression and other reasons.

A multicenter, cluster randomized controlled trial will be performed in all six psychiatric hospitals in Slovenia and will include twelve acute psychiatric wards. The trial will be prepared in accordance with the Consort guidelines.

The aims of the study are:

* To evaluate the effectiveness of verbal and non-verbal de-escalation techniques on the aggression incidence and severity.
* To evaluate the effectiveness of verbal and non-verbal de-escalation techniques on the incidence and duration of physical restraints.

Prior to the study, an information letter describing the study with a request to participate in the study will be sent to the professional managers in all psychiatric hospitals.

In Slovenia, six psychiatric hospitals provide inpatient psychiatric treatment. There are two acute psychiatric wards in each hospital, one for male and one for female patients. Subspecialized psychiatric wards, as the psychogeriatric ward, the acute psychiatric ward for adolescent and the acute forensic psychiatric ward will not be included.

We anticipate that approximately 6,000 subjects will be hospitalized in all twelve wards during the study.

The study will be conducted in two phases, a baseline period of five consecutive months and an intervention period during the same five consecutive months in the following year.

During the five months of the baseline period, the management of aggressive behavior in all psychiatric hospitals will be the same as usual. Before the five months of the intervention period, hospitals will be randomly assigned to either an experimental or control group in the 1:1 ratio. Randomization will be performed at the level of hospitals, not wards, to avoid possible transmission of the effect of the intervention among psychiatric hospital staff. The staff in the experimental group will receive training in verbal and nonverbal de-escalation techniques, and in the control group, the staff will manage aggressive behavior as usual. Regular annual training on the use of coercive measures will be conducted as usual in all hospitals.

The randomization will be performed after the baseline period, so the baseline data could not be biased. The hospital staff will be unaware of the aim and the design of the study. Psychiatric hospital managers will be informed that de-escalation training in all hospitals will be provided within 2 years.

The intervention will include training on verbal and nonverbal de-escalation techniques. The training will be prepared according to the recommendations of the Beta Project of the American Association for Emergency Psychiatry, the World Health Organization Quality Rights training to act, unite and empower for mental health and a handbook for the use of de-escalation skills in a hospital setting by Amdur E.

Data on aggressive incidents and the use of restraints will be obtained in the baseline and intervention phase. Aggressive incidents and severity will be measured using the Staff Observation Aggression Scale (SOAS-R). Data on physical restraints will be obtained from the standardized documentation required by the Mental Health Act, where the reason for the introduction is described (aggressive behavior, other reasons). Sociodemographic and clinical data of patients and data on bed capacities and the number of nursing staff will be summarized at the end of each study period from the hospital documentation and from medical records.

Data will be collected each month in all psychiatric hospitals. One of the staff members will be assigned to regularly remind the staff and to monitor the recording of incidents in each hospital. Data from SOAS-R forms and documentation for the use of physical restraint will be transferred to electronic databases by independent collaborators who are not familiar with the design of the study. All data will be anonymized The principal investigator and other researchers will regularly assess the compliance of the data collection with the protocol and verify the accuracy in relation to the source documents.

Protecting the benefits of the comparison group:

After the intervention period of the research, staff from the acute wards of psychiatric hospitals from the control group will receive de-escalation training.

Reasons for participant withdrawal from study:

Hospitals included in the study will be able to withdraw from the study at any time upon request.

Premature termination of study:

This study may be terminated prematurely if there is sufficient reasonable cause (insufficient compliance with protocol requirements and insufficiently complete data). Written notification, documenting the reason for study suspension, will be provided by the suspending party to investigator, funding agency and National Medical Ethics Committee.

Assessment of safety:

The principal investigator and collaborators from the psychiatric hospitals involved in the study will closely monitor the progress of the study to ensure the protection of human rights, the study to be conducted in accordance with the protocol and the quality and integrity of the study.

Ethics:

The study will be conducted in accordance with the principles of the World Medical Association Declaration of Helsinki, the Convention for the Protection of Human Rights and Dignity of the Human Being regarding the Application of Biology and Medicine and the Convention on Human Rights and Biomedicine. The study was approved from the National Medical Ethics Committee, Ministry of Health, Republic of Slovenia (0120-74/2018/).

Statistical analysis plan:

Primary outcomes: The incidence of aggressive events and restraint episodes will be presented as incident rates per 100 treatment days, with a 95% confidence interval. The incidence rate ratio (IRR) for an aggressive incident and physical restraint episodes between the experimental and control groups will be calculated for the baseline and intervention periods, then the change in IRR between the baseline and intervention period will be calculated. The difference in the incidence of aggression and restraints between the experimental and control groups will be tested using the Wald z-test. The effect of the intervention on the number of aggressive incidents and episodes of restraints, controlling for potential confounding patient characteristics will be examined using regression analyses.

Secondary outcomes: The severity of incidents will be measured using the SOAS-R scoring system, ranging from 0 to 22 points. The severity of aggressive incidents is defined categorically as the presence or the absence of a severe aggressive incident and numerically with the number of SOAS-R points. Incidents with a severity of nine or more points on the SOAS-R score will be regarded as severe incidents, as recommended by the authors of the SOAS-R (personal communication) and used in most research in recent years. The severity of aggressive incidents will be presented as the mean value of SOAS-R points, median and interquartile range. The difference in the severity of incidents between groups in each phase of the study will be calculated using the t-test or the Mann-Whitney U test. Differences in the duration of restraint episodes between the experimental and control groups will be presented by comparing the sum of restraint hours with the sum of treatment hours for all patients in each group and the study period. Then the risk ratios for the restraint hour between the experimental and control groups will be calculated for each study period.

The proportion of patients with at least one incident and then the risk ratio (RR) of aggression and restraints with 95% confidence interval in patients between the experimental and control groups will be calculated for the baseline and intervention period.

The characteristics of aggressive patients will be analyzed using descriptive statistical methods. For statistical analysis the IBM Statistical Package for the Social Sciences, version 25 and the Software environment for data analysis R will be used. The significance level of all statistical tests is determined at p < 0.05, two-sided.

ELIGIBILITY:
Inclusion Criteria:

* acute psychiatric ward - all patients, hospitalized during the study

Exclusion Criteria:

* acute psychogeriatric ward, acute psychiatric ward for adolescent, acute forensic psychiatric ward

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Number of aggressive incidents before and after the intervention. | Data for five months at baseline and for five months during the intervention period.
  Aggressive incidents will be measured using the SOAS-R scale. The number of aggressive incidents for the baseline period will be arranged according to which group the individual hospitals will be allocated to after randomization. The number of aggressive incidents will be calculated per 100 treatment days.
Number of physical restraint episodes before and after the intervention. | Data for five months at baseline and for five months during the intervention period.
  Data on restraint episodes will be obtained from the standardized documentation required by the Mental Health Act. The number of restraint episodes for the baseline period will be arranged according to which group the individual hospitals will be allocated to after randomization. The number of restraint episodes will be calculated per 100 treatment days.

SECONDARY OUTCOMES:
Severity of aggressive incidents before and after the intervention. | Data for five months at baseline and for five months during the intervention period.
  The severity of incidents will be measured using the SOAS-R scoring system, ranging from 0 to 22 points.
Duration of physical restraints episodes before and after the intervention. | Data for five months at baseline and for five months during the intervention period.
  The episode of physical restraint represents each individual restraint and covers the period from introduction to discontinuation. Data on duration of restraint episodes will be obtained from the standardized documentation required by the Mental Health Act.

OTHER OUTCOMES:
Proportion of aggressive patients before and after the intervention. | Data for five months at baseline and for five months during the intervention period.
  Data will be obtained from hospital registries and documentation.
Proportion of restraint patients before and after the intervention. | Data for five months at baseline and for five months during the intervention period.
  Data will be obtained from hospital registries and documentation.

CONTACTS AND LOCATIONS:
Overall Officials: Andreja Celofiga, Principal Investigator — University Medical Centre Maribor
Locations (6):
- Slovenia (6):
  - Psychiatric Hospital Begunje, Begunje na Gorenjskem
  - Psychiatric Hospital Idrija, Idrija
  - University Pychiatric Clinic Ljubljana, Ljubljana
  - Department of Psychiatry, University Medical Centre Maribor, Maribor
  - Psychiatric Hospital Ormoz, Ormož
  - Psychiatric Hospital Vojnik, Vojnik

IPD SHARING:
Plan to Share IPD: Yes
Data will be available on request, after data processing and publication of results.
Supporting Information: Study Protocol, CSR
Time Frame: Data will be available on request after data processing and publication of results (expected by the end of 2022).
Access Criteria: For research purposes.

REFERENCES:
- [Derived] Celofiga A, Kores Plesnicar B, Koprivsek J, Moskon M, Benkovic D, Gregoric Kumperscak H. Effectiveness of De-Escalation in Reducing Aggression and Coercion in Acute Psychiatric Units. A Cluster Randomized Study. Front Psychiatry. 2022 Apr 7;13:856153. doi: 10.3389/fpsyt.2022.856153. eCollection 2022. PMID 35463507